CLINICAL TRIAL: NCT04776070
Title: Establishing Malnutrition Diagnosis System by Using Artificial-intelligence Technology to Improve the Application of Clinical Pathway
Brief Title: Establishing Malnutrition Diagnosis System by Using Artificial-intelligence Technology
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Sichuan Academy of Medical Sciences (Other); Peking Union Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: JS-2768
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2021-02

CONDITIONS: Disease-related Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of malnutrition is estimated at 30-50% of hospitalized patients in China. Disease-related malnutrition increases the risk of infection, mortality, length of hospitalization as well as the economic burden. National Nutrition Plan proposed to reduce malnutrition, but a clear, effective roadmap and protocol has not existed yet. Several factors impede to resolve the above challenges. They include :1) the low efficiency of current malnutrition diagnosis methods; 2) the lack of dynamic, standard method that can evaluate nutritional status in quantitative way. To this end, the investigators aim to establish an artificial-intelligence malnutrition diagnosis system to improve the application of malnutrition Clinical Pathway. Firstly, the investigators will establish a multidimensional malnutrition large data set, based on our previously built national hospital nutrition screening data set.

It will contain deep 3D facial images, semi-structured and structured electronic medical record. Then, the investigators will use ensemble learning algorithm to establish a fully automatic, artificial-intelligence malnutrition diagnosis model that includes both etiological and phenotypic diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old);
* Within 48 hours of admission;
* Inpatients at high risk of malnutrition, such as malignant tumors, chronic obstructive pulmonary disease, etc;
* Han nationality;
* Able to given informed consent.

Exclusion Criteria:

* Patients with artificial facial changes (such as plastic surgery , head and neck radiotherapy , head and neck trauma);
* Diseases with special facial changes (such as acromegaly);
* High dose glucocorticoid users;
* Patients with facial edema;
* Emergency admission with an expected length of stay of less than 3 days;
* Other conditions researchers thought could not be included

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients in Peking Union Medical College
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-05-21 (Actual)

PRIMARY OUTCOMES:
malnutrition diagnosis | Within 48 hours of admission
  Using Global Leadership Initiative on Malnutrition(GLIM) to diagnose malnutrition among hospitalized patients

CONTACTS AND LOCATIONS:
Locations (1):
- Dongcheng district，Peking union medical college hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Sun MY, Wang Y, Zheng T, Wang X, Lin F, Zheng LY, Wang MY, Zhang PH, Chen LY, Yao Y, Sun J, Li ZN, Hu HY, Jiang H, Yue HY, Zhao Q, Wang HY, Han L, Ma X, Ji MT, Xu HX, Luo SY, Liu YH, Zhang Y, Han T, Li YS, Hou PP, Chen W. Health economic evaluation of an artificial intelligence (AI)-based rapid nutritional diagnostic system for hospitalised patients: A multicentre, randomised controlled trial. Clin Nutr. 2024 Oct;43(10):2327-2335. doi: 10.1016/j.clnu.2024.08.030. Epub 2024 Aug 30. PMID 39232261